CLINICAL TRIAL: NCT04944030
Title: Prediction in Silico of Therapeutic Response in a Prospective Cohort Study of Metastatic Lung Cancer Patients
Brief Title: Clinico-biological Data Collection Study of Metastatic Lung Cancer
Acronym: EPICURE_LUNG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICO-2020-19
Record Dates: First submitted 2021-06-15; First posted 2021-06-29 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Prospective clinico-biological database; Multi omic analysis; Prediction in silico
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Follow (Other): At each disease progression, patient will have specific interventions :
  * Metastasis biopsy
  * Biomarkers blood, urine and microbiota samples
  * Patient Reported Outcome (PRO)
  Interventions: Procedure: Metastasis biopsy

INTERVENTIONS:
Procedure: Metastasis biopsy — Metastasis biopsy will be performed for multi-omic analysis Biological/Vaccine: Biomarkers blood, urine and microbiota samples Biomarkers blood, urine and microbiota samples for multi-omic analysis Behavioral: Patient Reported Outcome (PRO) Patient Reported Outcome (PRO) will be collected throughout the study duration to assess quality of life, anxiety, depression distress, physical activity and food habits.

SUMMARY:
RATIONALE : Currently, the mechanisms associated with the response or resistance to treatment are poorly understood and are multifactorial. These mechanisms involve clinical and biological factors associated with the host and the tumor and possibly the patient's psycho-social environment.

PURPOSE : This trial will assess the use of a prospective database dedicated to patients with breast cancers that contains clinical data as well as epidemiological, psychological, emotional, social, imaging, biological and biopathological data. These data will allow a creation of new modelling algorithms in order to predict response and resistance to treatment.

DETAILED DESCRIPTION:
This prospective study will be conducted on first line metastatic lung cancer patients. Three phenotypic groups are identified on immunohistochemistry done at inclusion: on metastatic sites or lung tumor if local recurrence, usual treatment protocols are often guided by the following groups:

* For group 1: SCLC (small cell lung cancer)

  * Carbo or cisplatin + etoposide chemotherapy associated to atezolizumab or durvalumab
* For group 2: NSCLC (no small cell lung cancer) without oncogenic addiction:

  * Adenocarcinoma, NOS, sarcomatoïd carcinoma or large cell carcinoma with PDL1 expression level ≥ 50%: Carbo/cisplatin + pemetrexed + pembrolizumab or pembrolizumab alone.

In case of contra indication of pembrolizumab, treatment will be based on doublet of chemotherapy with platinum salt +/- bevacizumab - Adenocarcinoma, NOS, sarcomatoïde carcinoma or large cell carcinoma with PDL1 expression level < 50%: Carbo/cisplatin + pemetrexed + pembrolizumab.

In case of contra indication of pembrolizumab, treatment will be based on doublet of chemotherapy with platinum salt +/- bevacizumab

- Squamous cell carcinoma with PDL1 ≥ 50%: Carboplatin + paclitaxel + pembrolizumab or pembrolizumab alone.

In case of contra indication of pembrolizumab, treatment will be based on doublet of chemotherapy with platinum salt - Squamous cell carcinoma with PDL1 < 50%: Carboplatin + paclitaxel + pembrolizumab or pembrolizumab alone.

In case of contra indication of pembrolizumab, treatment will be based on doublet of chemotherapy with platinum salt

• For group 3: NSCLC NSCLC (no small cell lung cancerwith oncogenic addiction (KRAS G12c/BRAFV600E/NTRK/ROS1/ALK/EGFR/RET/NTRK/HER2):

* For which TKI is indicated: TKI as long as possible
* If TKI is not indicated: doublet of chemotherapy with platinum salt +/- pembrolizumab or pembrolizumab alone for PDL1 ≥ 50% or doublet of chemotherapy +/- bevacizumab

Further treatment lines are administered according to standard practice. Biological and histological assessments are performed on specific metastasis biopsy samples done at baseline and at each progression.

Physical exam, standard laboratory tests, imaging (CT (computerized tomography) scan, PET-CT (Positron emission tomography-computed tomography) and bone scan (for patients with bone metastasis) will be performed every 2 to 3 months according to patient group. Clinical, biological, pathological, epidemiological, socio-economic and multiomic data will be collected throughout the study duration. These massive data will be used to create new algorithms in order to help clinicians to predict treatment response

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening biopsy, blood sample and questionnaires
* 18 years old at time of written consent
* Patient with histologically confirmed lung cancer
* Lung cancer metastatic disease or locally advanced not eligible for local curative treatment intent
* Performance status ≤ 2 (according to WHO criteria)
* Indication of any systemic therapeutic strategy can be performed alongside this current cohort in accordance with national and / or international recommendations.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Patient must be affiliated to a Social Health Insurance

Exclusion Criteria:

* Other malignancy treated within the last 3 years (except non-melanoma skin cancer or in situ carcinoma of the cervix)
* Other neuroendocrine tumour than small cell or large cell carcinoma.
* Pregnant or nursing patient
* Individual deprived of liberty or placed under the authority of a tutor
* Impossibility to submit to the medical follow-up of this clinical trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 15 years
  Overall Survival is defined by the delay between the date of inclusion and the date of death or last follow-up assessment

SECONDARY OUTCOMES:
To describe response to treatment for each therapeutic sequence | 15 years
  The response to treatment will be assessed using local radiological review according to RECIST 1.1 criteria
To evaluate progression free survival (PFS) for each therapeutic sequence | 15 years
  Progression Free survival is defined by the delay between the first dose of a treatment sequence and the date of documented disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: JUDITH RAIMBOURG, MD,PHD, Principal Investigator — judith.raimbourg@ico.unicancer.fr
Locations (2):
- France (2):
  - Institut de Cancerologie de L'Ouest, Angers
  - Institut de Cancerologie de L'Ouest, Saint-Herblain